CLINICAL TRIAL: NCT06210412
Title: The Effect of Health Education and Yoga Practices Given According to Pender's Health Promotion Model on Menopausal Symptoms and Quality of Life: A Randomized Controlled Study
Brief Title: The Effect of Health Education and Yoga on Menopause Symptoms and Quality of Life According to Pender's Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Meltem Altınışık, Senior instructor, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ETK00-2023-0262
Record Dates: First submitted 2024-01-05; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Quality of Life; Health Education; Yoga; Menopause Symptoms
Keywords: Menopause symptoms; health education; yoga; quality of life
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Intervention Model Description: The introductory information form and MÖYKÖ tests will be applied. Women with high MÖYKÖ scores will be divided into experimental and control groups using purposeful sampling, according to the lottery method, and those in the experimental group will be contacted by phone and asked to come to the Famagusta Development Academy (MGA) on the day and time determined. Sessions will begin after 12 weeks of health training and Hatha yoga practice are planned. At the end of 12 weeks, final tests will be administered to women who have participated for at least 10 weeks. Those in the control group will be called by phone and invited to MGA Maraş for their first test, and an appointment will be made 12 weeks later for their final test.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- health education and yoga intervention group (Experimental): Health education program based on the Penderin Health Promotion Model; It consists of 10 sessions as a program focused on the management of menopause (increasing the quality of life by teaching physical, psychological and social coping methods in menopause, yoga practices and their importance). In the first week, introduction, first tests (Sociodemographic data form, MÖYKÖ), and general introduction of the program will be made. It is a program in which active education methods (question and answer, role play, demonstration, etc.) are used, with each session planned to last approximately 30 minutes. Final tests will be performed at the end of 12 weeks.
  Yoga practice will be carried out as 45-minute sessions 2 days a week, which will last for 12 weeks, following the health education program.12. At the end of the week, MOQÖ and Yoga Transformation Impact Scale will be applied to those who have completed 10 weeks.
  Interventions: Behavioral: health education and yoga intervention group
- Control group (No Intervention): Voluntary consent forms, which will be informed during the interview, and a sociodemographic data form, Menopause-Specific Quality of Life Scale, will be filled in by participants who wish to participate in the research. They will then be invited to undergo final testing after 12 weeks.

INTERVENTIONS:
Behavioral: health education and yoga intervention group — Health education program based on the Penderin Health Promotion Model; It consists of 10 sessions as a program focused on the management of menopause (increasing the quality of life by teaching physical, psychological and social coping methods in menopause, yoga practices and their importance). In the first week, introduction, first tests (Sociodemographic data form, MÖYKÖ), and general introduction of the program will be made. It is a program in which active education methods (question and answer, role play, demonstration, etc.) are used, with each session planned to last approximately 30 minutes. Final tests will be performed at the end of 12 weeks.
  Yoga practice will be carried out as 45-minute sessions 2 days a week, which will last for 12 weeks, following the health education program.12. At the end of the week, MOQÖ and Yoga Transformation Impact Scale will be applied to those who have completed 10 weeks.
  Arms: health education and yoga intervention group

SUMMARY:
The aim of the study is to examine the effect of health education and yoga intervention prepared according to Pender's Health Promotion Model on menopausal women's "menopause-specific quality of life" compared to routine care. Health education and yoga will be conducted by a certified and responsible investigator. After obtaining informed consent from the participants, the scales will be applied before and after health education and yoga practice.

DETAILED DESCRIPTION:
It is known that the symptoms experienced by women during menopause affect the woman's quality of life. Many methods have been used in the literature to manage menopause symptoms. However, this study is important to present health education prepared according to Pender's health development model, which will enable women to develop health responsibility awareness, and to manage and alleviate menopausal symptoms of yoga practice planned in this context, to determine its effect on quality of life and to provide a source for literature.

Research hypotheses:

H0= There is no difference between menopause-specific quality of life score averages.

H1= There is a difference between menopause-specific quality of life score averages.

Research question:

1.What are the yoga transformation effect scale scores of the participants in the experimental group after the yoga intervention?

Data Collection Tools Three data collection forms will be used in the research. There is an Introductory Information Form, "Menopause-Specific Quality of Life Scale", and "Yoga Transformation Scale".

ELIGIBILITY:
Inclusion Criteria:

* Been in menopause for at least 1 year and at most 5 years
* Experiencing menopausal symptoms at least 3 to 4 times a week in the last 3 months
* Those who have no physical disability to practice yoga
* Able to speak and understand Turkish

Exclusion Criteria:

* Those who receive hormone replacement therapy
* Those who have undergone surgical menopause
* Having done yoga before

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — menopause womans
Enrollment: 66 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
The Effect of Health Education and Yoga on Menopause-Specific Quality of Life in Women | 12 week
  Menopause-Specific Quality of Life Scale-MSQS "Menopause-Specific Quality of Life Scale (MSQQ)" The Turkish validity and reliability of the scale developed by Hilditch et al. in 1996 was tested by Kharbouch and Şahin in 2005. Made by. The scale consists of four domains: vasomotor, psychosocial, physical and sexual, contains 29 Likert-type statements, and as the score obtained from the scale increases, the severity of the complaint increases and the quality of life decreases. Since the average score is used in the total scale, the lowest score that can be obtained from the scale is 0 and the highest score is 6. Sub-domains of the scale; It consists of four subdomains: vasomotor (questions 1-3), psychosocial (questions 4-10), physical (questions 11-26) and sexual (questions 27-29). E-mail permission was obtained for the use of the scale (32).

SECONDARY OUTCOMES:
Determining the effect of Health Education and Yoga on the "Yoga Transformation Effect Scale" in Menopausal Women | 12 Weeks
  Birdee et al. (2015), the Turkish reliability and validity study was conducted by Tetik Küçükelçi (2018). The scale consists of 11 items and three subscales: body (4 items), breath (4 items) and mind (3 items); It measures individuals' yoga self-efficacy levels. An increase in the score obtained from the scale subscale scores indicates a high yoga-self-efficacy status. The Cronbach's alpha value of the scale was 0.88 in the original study; In the current study, it was found to be 0.95 (31). E-mail permission was obtained for the use of the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Altınışık, Principal Investigator — eastern meditternean ünivercity
Locations (1):
- Meltem Altınışık, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, ICF, CSR

REFERENCES:
- [Result] Lambiase MJ, Thurston RC. Physical activity and sleep among midlife women with vasomotor symptoms. Menopause. 2013 Sep;20(9):946-52. doi: 10.1097/GME.0b013e3182844110. PMID 23531686
- [Result] Jones SM, Guthrie KA, Reed SD, Landis CA, Sternfeld B, LaCroix AZ, Dunn A, Burr RL, Newton KM. A yoga & exercise randomized controlled trial for vasomotor symptoms: Effects on heart rate variability. Complement Ther Med. 2016 Jun;26:66-71. doi: 10.1016/j.ctim.2016.03.001. Epub 2016 Mar 4. PMID 27261984
- [Result] Kimura N, Nagata N. The requirement of guanine nucleotides for glucagon stimulation of adenylate cyclase in rat liver plasma membranes. J Biol Chem. 1977 Jun 10;252(11):3829-35. No abstract available. PMID 863905
- [Result] Kaminetzky H. Sodium in pregnancy: part I. Ariz Med. 1978 Apr;35(4):255-6. No abstract available. PMID 655871